CLINICAL TRIAL: NCT04700098
Title: Enhancing Pulmonary Rehabilitation in Veterans With Chronic Obstructive Pulmonary Disease Through Internet-based Cognitive-behavioral Treatment for Insomnia
Brief Title: Internet-based Cognitive-behavioral Treatment for Insomnia in COPD Patients Undergoing Pulmonary Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F3513-R
Record Dates: First submitted 2021-01-04; First posted 2021-01-07 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; Insomnia
Keywords: Chronic Obstructive Pulmonary Disease; Insomnia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Individuals will be assigned to either an internet-based behavioral treatment for insomnia or online insomnia patient education.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Internet-based behavioral treatment for insomnia (Experimental): Internet version of cognitive-behavioral treatment for insomnia
  Interventions: Behavioral: Internet-based behavioral treatment for insomnia
- Online insomnia patient education (Experimental): Online insomnia patient education
  Interventions: Behavioral: Online insomnia patient education

INTERVENTIONS:
Behavioral: Internet-based behavioral treatment for insomnia — Internet version of cognitive-behavioral treatment for insomnia
  Arms: Internet-based behavioral treatment for insomnia
Behavioral: Online insomnia patient education — Online insomnia patient education
  Arms: Online insomnia patient education

SUMMARY:
This study is a randomized controlled trial (RCT) to compare sleep and health-related functioning in Veterans with chronic obstructive pulmonary disease (COPD) and insomnia receiving an Internet-based behavioral treatment for insomnia versus online insomnia patient education. Participants will undergo a sleep and health assessment that will be performed at baseline, post-treatment, and 3-months later. Participants will be randomly assigned to either Internet-based behavioral treatment for insomnia or online insomnia patient education.

DETAILED DESCRIPTION:
Veterans with chronic obstructive pulmonary disease (COPD) are a vulnerable group for developing insomnia. Insomnia has been found to be associated with limitations in activities of daily living (ADL), lower physical activity levels, poor quality of life, greater COPD symptom severity, and reduced exercise performance. Cognitive-behavioral therapy for insomnia (CBT-I) is an efficacious and durable non-pharmacological treatment for insomnia that provides guidance on changing unhealthy sleep-related beliefs and behaviors across a variety of illnesses. CBT-I not only improves sleep-specific symptoms of insomnia but also improves quality of life and daytime function, reduces ADL limitations, and improves condition-specific symptoms.

This study is a randomized controlled trial (RCT) to compare sleep and health-related functioning in Veterans with chronic obstructive pulmonary disease (COPD) and insomnia receiving an Internet-based behavioral treatment for insomnia versus online insomnia patient education. Veterans 40 years and older, who received care from the VA Pittsburgh Healthcare System, and who have COPD and insomnia will be recruited for this study. Participants will undergo a sleep and health assessment that will be performed at baseline, post-treatment, and 3-months later. Participants will be randomly assigned to either Internet-based behavioral treatment for insomnia or online insomnia patient education. Both the insomnia treatment and patient education will be provided remotely.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years and older
* Primary diagnosis of COPD defined by GOLD
* Meets criteria for Insomnia Disorder
* At least moderate insomnia severity based on Insomnia Severity Index score >7
* Stable psychiatric and medical conditions
* Must have telephone, email, and reliable Internet access via computer, smartphone, or tablet

Exclusion Criteria:

* Untreated current major depression
* Serious suicidal risk
* Substance abuse disorder within past 3 months
* History of bipolar or psychosis
* Untreated restless legs syndrome, delayed sleep phase syndrome, irregular sleep schedules
* Very severe untreated obstructive sleep apnea
* Severe excessive daytime sleepiness based on Epworth Sleepiness Scale score > 16
* Restrictive lung disease (FEV1/FVC 70 and FEV1 < 80% predicted) or asthma
* Plans to move during the following 6 months
* Non-English speaking or sensory deficits

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | Baseline to post-treatment and 3-months post-treatment
  The Insomnia Severity Index is a 7-item self-report questionnaire assessing nature, severity and impact of insomnia symptoms. The total score ranges from 0 to 28, with higher scores indicating worse insomnia severity.
St. George's Respiratory Questionnaire | 6-months post-pulmonary rehabilitation
  The SGRQ is a 50-item measure assessing disease-specific quality of life. The total SGRQ score, which reflects the overall impact of the disease on quality of life, ranges from 0 to 100, with higher scores indicating greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Faith S Luyster, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (2):
- United States (2):
  - John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT04700098/ICF_000.pdf